CLINICAL TRIAL: NCT06235723
Title: Impact of Virtual Reality on Peri-interventional Pain, Anxiety and Distress in a Pediatric Oncology Outpatient Clinic: a Randomized Controlled Trial
Brief Title: Impact of Virtual Reality on Peri-interventional Pain, Anxiety and Distress in a Pediatric Oncology Outpatient Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: VirtualReality2023
Record Dates: First submitted 2023-12-23; First posted 2024-02-01 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Pediatric Cancer; Procedural Anxiety; Procedural Pain
Keywords: Virtual Reality; Pediatric Oncoloy; Outpatient Clinic; Peri-interventional Pain
MeSH Terms: conditions — Neoplasms; Pain, Procedural

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOC (A) (No Intervention): SOC = Standard-of-Care
- VR (B) (Experimental): VR = Virtual Reality
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Virtual Reality was used before and during punctures. For every observation patients underwent either port puncture or peripheral venous puncture. One examination was carried out according to the Standard-of-Care. The other one was carried out with the additional use of VR. Participants watched a passive distraction video.
  Arms: VR (B)

SUMMARY:
Pain and anxiety-inducing interventions have a major impact on pediatric patients. Pain reduction by virtual reality (VR) during port and vein punctures is well studied. This study investigates peri-interventional reduction of pain, anxiety and distress using VR compared to the standard of care (SOC) in a pediatric oncology outpatient clinic.

In a randomized, controlled cross-over design, patients aged 6-18 years experience potentially painful interventions accompanied by VR. All patients included in the study underwent port puncture or peripheral venous puncture in two observations : SOC (A) and VR (B) in a randomized order. Observational instruments include Numeral Rating Scale (NRS), Faces Pain Scale revised (FPS-r), Behavioral Approach Avoidance Distress Scale (BAADS), modified Yale Preoperative Anxiety Scale (mYPAS-SF). In addition, parents and staff are interviewed. Specific conditions for VR in an outpatient clinic setting are being discussed.

ELIGIBILITY:
Inclusion Criteria:

* aged 6-18 years
* any sex
* port puncture or placement of a peripheral venous catheter in pediatric outpatient clinic
* hematological or oncological diagnosis
* informed consent

Exclusion Criteria:

* epilepsy
* coronary artery disease
* history of severe vertigo
* obstacles to putting on and wearing VR glasses
* lack of informed consent for study participation.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Procedural Pain measured with Numeric Rating Scale (NRS; scale 0-10; higher score stating higher levels of pain) | pre-, peri-, post-interventional (before puncture when entering intervention room, during puncture and 5 minutes after puncture)
  Virtual Reality vs. Standard-of-Care
Procedural Anxiety measured with modified Yale Preoperative Anxiety Scale (mYPAS-SF; scale 23-100; higher score stating higher levels of anxiety) | pre-, peri-interventional (before puncture when entering intervention room and during puncture)
  Virtual Reality vs. Standard-of-Care
Procedural Distress measured with Behavioral Approach Avoidance Distress Scale (BAADS; scale 0-10; higher score stating higher levels of distress) | pre-, peri-interventional (before puncture when entering intervention room and during puncture)
  Virtual Reality vs. Standard-of-Care

SECONDARY OUTCOMES:
Acceptance of VR in pediatric procedures (questionnaire using a 5-point-likert-scale) | post-interventional (immediately after the intervention)
  Parents and patients were given different statements
Implementation factors for VR in pediatric outpatient clinics (qualitive questionnaire) | through study completion, ~ 1.5 years in total
  Involved staff were asked about experience/feedback

CONTACTS AND LOCATIONS:
Overall Officials: Urs Mücke, Dr., Principal Investigator — Hannover Medical School
Locations (1):
- Medical School Hanover, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reitze A, Voigt M, Klawonn F, Dusch M, Grigull L, Mucke U. Impact of virtual reality on peri-interventional pain, anxiety and distress in a pediatric oncology outpatient clinic: a randomized controlled trial. BMC Pediatr. 2024 Aug 3;24(1):501. doi: 10.1186/s12887-024-04952-3. PMID 39097718